CLINICAL TRIAL: NCT00845481
Title: A Plaque Test Comparing 4 Steroids With Daivobet® Ointment and a Vehicle Control for the Treatment of Psoriasis Vulgaris
Brief Title: A Plaque Test Comparing the Anti-psoriatic Effect of Marketed Products for Topical Use for Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: PLQ-002
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients apply all products (Experimental)
  Interventions: Drug: Daivobet® ointment; Drug: Betnovat® ointment; Drug: Diprosalic ointment; Drug: Dermovat ointment; Drug: Elocon ointment; Drug: Daivobet® ointment vehicle

INTERVENTIONS:
Drug: Daivobet® ointment — Once daily application 6 days a week for 3 weeks
Drug: Betnovat® ointment — Once daily application 6 days a week for 3 weeks
Drug: Diprosalic ointment — Once daily application 6 days a week for 3 weeks
Drug: Dermovat ointment — Once daily application 6 days a week for 3 weeks
Drug: Elocon ointment — Once daily application 6 days a week for 3 weeks
Drug: Daivobet® ointment vehicle — Once daily application 6 days a week for 3 weeks

SUMMARY:
The purpose of the study is to compare the anti-psoriatic effect of marketed products with Daivobet® ointment in a plaque test

ELIGIBILITY:
Inclusion Criteria: (in summary)

* Subjects having understood and signed an informed consent form
* All skin types
* Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms, legs or trunk. The lesions must have a total size suitable for application. The subjects should be asked if their lesions have been stable
* Subjects willing and able to follow all the study procedures and complete the whole study
* Subjects affiliated to social security system

Exclusion Criteria: (in summary)

* Females who are pregnant, of child-bearing potential and who wish to become pregnant during the study, or who are breast feeding
* Subjects using biological therapies (marketed or not marketed) with a possible effect on psoriasis (e.g. alefacept, efalizumab, etanercept, infliximab, adalimumab) within 12 weeks prior to study drug administration
* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D-analogues, retinoids, immunosuppressants) within the 4-week period prior to randomisation
* Subjects using one of the following topical drugs for the treatment of psoriasis within four (4) weeks prior to study drug administration: - Potent or very potent (WHO group III-IV) corticosteroids - PUVA or Grenz ray therapy
* Subjects using one of the following topical drugs for the treatment of psoriasis within two (2) weeks prior to study drug administration: - WHO group I-II corticosteroids - Topical retinoids - Vitamin D-analogues - Topical immunomodulators (e.g. macrolides) - Anthracen derivatives - Tar - Salicylic acid - UVB therapy
* Subjects with skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds within the plaque test areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Pharma Investigational Site, Saint Quentin Yvelines Cedex, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated: Treatments are given at the same time on different locations of the skin with psoriasis in the same group of participants.
Period: Overall Study
Arm/Group | Patients Treated
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (9.6)
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 67 years | 23
  >=68 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Region of Enrollment [Number; unit: participants]
  France | 24

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Change in Total Clinical Score (TCS) at End of Treatment Compared to Baseline for Daivobet® Ointment
Description: The Total Clinical Score is the sum of three psoriasis scores (redness, thickness, and scaliness) and will range from 0 (best) to 9 (worst)
Time Frame: Baseline and 3 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Patients Treated With Daivobet® Ointment: Treatments are given at the same time on different locations of the skin with psoriasis in the same group of participants. The treatment for this outcome measure is Daivobet® ointment
Arm/Group | Patients Treated With Daivobet® Ointment
Number analyzed (Participants) | 24
Scores on a scale | -5.15 (1.31)

2. Primary Outcome: The Absolute Change in Total Clinical Score (TCS) at End of Treatment Compared to Baseline for Betnovat® Ointment
Description: as for outcome 1
Time Frame: Baseline and 3 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Patients Treated With Betnovat® Ointment: Treatments are given at the same time on different locations of the skin with psoriasis in the same group of participants. The treatment for this outcome measure is Betnovat® ointment
Arm/Group | Patients Treated With Betnovat® Ointment
Number analyzed (Participants) | 24
Scores on a scale | -3.33 (2.44)

3. Primary Outcome: The Absolute Change in Total Clinical Score (TCS) at End of Treatment Compared to Baseline for Elocon Ointment
Description: as for outcome 1
Time Frame: Baseline and 3 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Patients Treated With Elocon Ointment: Treatments are given at the same time on different locations of the skin with psoriasis in the same group of participants. The treatment for this outcome measure is Elocon ointment
Arm/Group | Patients Treated With Elocon Ointment
Number analyzed (Participants) | 24
Scores on a scale | -4.50 (1.74)

4. Primary Outcome: The Absolute Change in Total Clinical Score (TCS) at End of Treatment Compared to Baseline for Daivobet Ointment Vehicle
Description: as for outcome 1
Time Frame: Baseline and 3 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Patients Treated With Daivobet® Ointment Vehicle: Treatments are given at the same time on different locations of the skin with psoriasis in the same group of participants. The treatment for this outcome measure is Daivobet® Ointment vehicle
Arm/Group | Patients Treated With Daivobet® Ointment Vehicle
Number analyzed (Participants) | 24
Scores on a scale | -1.91 (1.15)

5. Primary Outcome: The Absolute Change in Total Clinical Score (TCS) at End of Treatment Compared to Baseline for Dermovat Ointment
Description: as for outcome 1
Time Frame: Baseline and 3 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Patients Treated With Dermovat Ointment: Treatments are given at the same time on different locations of the skin with psoriasis in the same group of participants. The treatment for this outcome measure is Dermovat ointment
Arm/Group | Patients Treated With Dermovat Ointment
Number analyzed (Participants) | 24
Scores on a scale | -5.71 (1.39)

6. Primary Outcome: The Absolute Change in Total Clinical Score (TCS) at End of Treatment Compared to Baseline for Diprosalic Ointment
Description: as for outcome 1
Time Frame: Baseline and 3 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Patients Treated With Diprosalic Ointment: Treatments are given at the same time on different locations of the skin with psoriasis in the same group of participants. The treatment for this outcome measure is Diprosalic ointment
Arm/Group | Patients Treated With Diprosalic Ointment
Number analyzed (Participants) | 24
Scores on a scale | -4.50 (1.84)

ADVERSE EVENTS:
Arm/Group | Patients Treated
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO retains the right to publish the results of this clinical trial